CLINICAL TRIAL: NCT05099315
Title: Identification of Skin-associated Microbiota in Atopic Dermatitis Patients Undergoing Systemic Therapy
Brief Title: Microbiome in Atopic Dermatitis Under Systemic Therapy
Acronym: BIO-AD
Status: Recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Margitta Worm, Prof. Dr. med. Margitta Worm, Charite University, Berlin, Germany
Other Study IDs: Microbiome and AD
Record Dates: First submitted 2021-07-20; First posted 2021-10-29 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Atopic Dermatitis
Keywords: dupilumab; cyclosporine; skin microbiome; baricitinib
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — 1. Serum,
  2. Peripheral blood mononuclear cells
  3. Skin swab for microbiome analysis
  4. Genetic examination of the filaggringen mutation status
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Dupilumab treated Patients (observational): Patients with atopic dermatitis with indication for dupilumab treatment will be observed.
  Interventions: Other: not applicable, observational study
- Cyclosporine treated Patients (observational): Patients with atopic dermatitis with indication for cyclosporine treatment will be observed.
  Interventions: Other: not applicable, observational study
- Baricitinib treated Patients (observational): Patients with atopic dermatitis with indication for baricitinib treatment will be observed.
  Interventions: Other: not applicable, observational study

INTERVENTIONS:
Other: not applicable, observational study — Patients undergoing systemic therapy according to international accepted guidelines for the therapy of atopic dermatitis, observational study

SUMMARY:
The skin microbiome plays a role in the pathogenesis of atopic dermatitis. However, it is unclear whether the range of microbiota on the skin is the cause or consequence of atopic skin inflammation.

The influence of new systemic therapies for the treatment of moderate to severe atopic dermatitis (such as biologics or Janus kinase inhibitors) on the skin microbiome is largely unknown.

The main aim of this scientific exploratory study is to investigate whether and how the skin microbiome changes in patients with moderate to severe atopic dermatitis during systemic therapy. This not only allows new hypotheses to be generated on the pathogenesis of atopic dermatitis, but also new objective scales for the severity of atopic dermatitis can be developed.

DETAILED DESCRIPTION:
A better understanding of the pathology of atopic dermatitis could lead to the development of new therapeutic strategies for this disease and contribute to better and more targeted disease management - an advantage for all patients with atopic dermatitis.

The routine examinations are carried out every quarter with routine visits over two years. The dates before, 6, 12, and 24 months after the initiation of systemic therapy are relevant for this study. Deviations from normal practice are not intended.

Patients in whom a new initiation of systemic therapy is planned will be invited for a follow-up 6 weeks after initiation and quarterly follow-up visits.

Blood samples must be obtained for the examination. The blood is taken to determine the systemic level of inflammatory mediators (serological biomarkers, PBMCs) and for genetic examinations (e.g. filaggrin gene mutation - FLG) as well as mRNA / lncRNA profile. The skin physiological examinations are not invasive or pain-related procedures. Microbiome sampling will be conducted by a skin swab of the inter-scapular region.

The blood / skin samples taken as part of this scientific study are pseudonymized in the research laboratories. The samples are stored in the laboratories for a period of 5 years after the end of the study and then destroyed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe atopic dermatitis
* Indication for systemic therapy

Exclusion Criteria:

* Patients under 18 years of age upon introducing systemic therapy
* Pregnant and lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with moderate to severe atopic dermatitis presenting in the clinic of Dermatology, Charité - Universitätsmedizin Berlin, Germany.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of the microbial composition | 1 year
  Comparison of the microbial composition of the skin before, 6 and 12 months after the initiation of systemic therapy.
Comparison of microbial composition of the skin with serological biomarkers | 1 year
  Comparison of microbial composition of the skin with serological biomarkers (z.B.TARC, TSLP, CCL27).

SECONDARY OUTCOMES:
Microbial composition and skin barrier function | 1 year
  Comparison of the microbial composition of the skin with the skin physiology (including transepidermal water loss, sebumetry)
Correlation of main microbial representants of skin microbiome | 1 year
  Correlation of the S. aureus to the P. acnes ratio
Correlation of microbiome and severity of atopic dermatitis EASI | 2 years
  Correlation of the microbiome with the Eczema Area and Severity Index (EASI). EASI ranges from 0-72, increasing severity with increasing score.
Correlation of microbiome and severity of atopic dermatitis SCORAD | 2 years
  Correlation of the microbiome with Scoring of Atopic Dermatitis (SCORAD). SCORAD ranges from 0-103, increasing severity with increasing score.
Association of the skin microbiome with the mRNA EASI | 2 years
  Correlation of the main representants of skin microbiota and the Eczema Area and Severity Index (EASI). EASI ranges from 0-72, increasing severity with increasing score.
Association of the skin microbiome with the mRNA SCORAD | 2 years
  Correlation of the main representants of skin microbiota and Scoring of Atopic Dermatitis (SCORAD). SCORAD ranges from 0-103, increasing severity with increasing score.

CONTACTS AND LOCATIONS:
Locations (1):
- Dpt of Dermatology and Allergology, Charité - Universitätsmedizin Berlin, Berlin, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided